CLINICAL TRIAL: NCT03286322
Title: Comparison of a Classical Rehabilitation Method and a Specific Rehabilitation Method of the Cervical Spine to Improve Balance in Elderly Patients
Brief Title: Comparison of a Classical Rehabilitation Method and a Specific Rehabilitation Method of the Cervical Spine
Acronym: SATRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00521-50
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Loss of Balance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy cervical spine (Experimental)
  Interventions: Other: manuel therapy cervical spine
- control group (Sham Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: manuel therapy cervical spine — the manuel therapy in physiotherapy is focused on the cervival spine
  Arms: manual therapy cervical spine
Other: control group — the manuel therapy in physiotherapy is classic and not focused on the cervival spine
  Arms: control group

SUMMARY:
In more than 90% of cases, victims of fall are elderly people over 65. Nearly the third of those people fall at least 1 time by year. The incidence substantially increases for people over 80 and women are at higher risk than men.

The value of balance rehabilitation no longer needs to be demonstrated in Gerontology. Nevertheless, a more specific therapy based on the aged-related cervical problems seems to be essential. Indeed, those problems are numerous (arthrosis-like pains, joint stiffness, muscular contractures…) and often lessen vestibular and/or proprioceptive afferents. The cervical spine is a link between different systems which regulate balance, as the visual, vestibular and cervical systems (muscular, articular afferents…), and this role is key to balance control. Indeed, the cervical spine owns an exceptional function thanks to Ruffinian corpuscles, muscle and neurotendinal spindles.

Many studies point up the importance of the relation between balance, cervical spine and vestibular system, and others between tissue changes and postural adaptations in elderly people. Nevertheless, the take into consideration of all these data and their impacts in rehabilitation has not been reported yet.

This brings us to question the added-value of a cervical mobility management in balance rehabilitation in Gerontology.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 hospitalized in rehabilitation department and long-term unit of Cimiez Hospital
* With MMSE > 20
* In need of balance rehabilitation
* Who can stand Bipodal position for >1 minute
* Who can walk for more than 10 meters without walking aid
* Having signed an informed consent
* Affiliated to a health insurance plan

Exclusion Criteria:

* Motor neurological deficit, specific vestibular pathologies
* Patient hospitalized for traumatological pathology or who has been hospitalized for traumatological pathology within 3 months
* Vulnerable people: adults under guardianship, deprived of freedom

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-12-16 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage decrease of the wobbling surface eyes open on steady ground, on a posturology platform | at 3 weeks
  To compare the balance improvement, thanks to a posturology platform, between 2 groups of elderly patients hospitalized for balance disorders, in order to highlight the way of manual therapy in physiotherapy, focused on the cervical spine, can increase these parameters and contribute to lessen the risk of falls in elderly people.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GONFRIER, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France